CLINICAL TRIAL: NCT00559156
Title: Phase 2 Study Assessing the Impact of Parenteral Administration of the Immunomodulater Oral IMPACT® for Postoperative Radiochemotherapy in Patients With Carcinoma of the Head and Neck
Brief Title: Arginine/Omega-3 Fatty Acids/Nucleotides Nutritional Supplement in Treating Patients With Stage III or Stage IV Head and Neck Cancer Undergoing Chemotherapy and Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574125; CLCC-IMPACT-RT; INCA-RECF0286
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Arginine; Cisplatin; Chemotherapy, Adjuvant; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Oral Impact Product
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oral Impact (Experimental): Oral Impact Supplement: 3 bags/day, 5 days before each chemotherapy
  Interventions: Dietary Supplement: arginine/omega-3 fatty acids/nucleotides oral supplement; Drug: cisplatin; Procedure: adjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Dietary Supplement: arginine/omega-3 fatty acids/nucleotides oral supplement
  Other Names: Oral Impact
Drug: cisplatin
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving a nutritional supplement containing arginine, omega-3 fatty acids, and nucleotides to patients undergoing chemotherapy and radiation therapy may stimulate the immune system and help the body build a stronger immune response.

PURPOSE: This phase II trial is studying how well an arginine/omega-3 fatty acids/nucleotides nutritional supplement works in treating patients with stage III or stage IV head and neck cancer undergoing chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the effects of immunomodulator arginine/omega-3 fatty acids/nucleotides oral supplement (Oral IMPACT®) administered via percutaneous gastrostomy during adjuvant chemoradiotherapy in patients with stage III or IV epidermoid head and neck cancer.

OUTLINE: This is a multicenter study.

Patients undergo radiotherapy 5 days a week for 6½ weeks. Patients receive cisplatin IV during weeks 1, 4, and 7 of radiotherapy. Patients also receive arginine/omega-3 fatty acids/nucleotides oral supplement (Oral IMPACT®) via percutaneous gastrostomy tube 3 times daily for 5 days before each chemotherapy treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of head and neck cancer meeting the following criteria:

  * Epidermoid carcinoma
  * Stage III or IV disease
* Must have percutaneous gastrostomy tube in place
* Must have undergone prior surgery for head and neck cancer within the past 6-8 weeks
* No cerebral metastases

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* WBC > 4,000/mm³
* ANC > 2,000/mm³
* Platelet count > 100,000/mm³
* PTT ≥ 50%
* Creatinine < 130 μmol/L
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No severe sepsis
* No requirement for parenteral nutrition
* No pre-existing digestive pathology that results in bowel obstruction, nausea, vomiting, and/or abdominal pain > grade 1

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Effects of immunomodulator arginine/omega-3 fatty acids/nucleotides oral supplement (Oral IMPACT®) administered via percutaneous gastrostomy during adjuvant chemoradiotherapy | 90 days after radiotherapy
  Toxicities grades 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Senesse, MD, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle